CLINICAL TRIAL: NCT01960621
Title: The Effect of Cyclodextrin on Sensory Nerve Activity and the Cough Relex in Man: A Novel Anti-Tussive Therapy
Brief Title: Effect of Cyclodextrin on Sensory Nerve Activity: A Novel Anti-tussive Therapy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study has not been able to start due to difficulty in obtaining an intravenous formulation of cyclodextrin (intravenous 2HPBCD) suitable for man
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 06/Q0406/102
Record Dates: First submitted 2008-05-08; First posted 2013-10-10 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Cough
MeSH Terms: conditions — Cough | interventions — Cyclodextrins

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- 2 (Experimental)
  Interventions: Drug: cyclodextrin

INTERVENTIONS:
Drug: cyclodextrin — intravenous

SUMMARY:
The investigators want to see whether the test drug in this research study, 2-hydroxypropyl-beta-cyclodextrin (2HPBCD), might potentially be able to improve cough in healthy volunteers. The investigators are initially recruiting healthy volunteers such as who are free from any respiratory disease and not on any concurrent medication, so there are no confusing effects from pre-existing respiratory symptoms or disease, nor interaction of any medication with the test drug.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-smoking participants (we have excluded smoking participants in light of the greater potential for cough to be present as a result of their smoking habit and they may be unduly sensitive to inhaled cough stimuli, such as the inhaled capsaicin cough challenge)
* Age 18-65 years
* No history of respiratory disease
* Normal baseline spirometry as predicted for age, sex and height (we have excluded those with abnormal spirometry, as we aim to induce cough in our otherwise healthy volunteer participants. Also, abnormal spirometry in the presence of no respiratory symptoms - may indicate an underlying lung condition that needs attention, and such participants will be told their result and with their consent, the information will be forwarded to their General Practitioner, as part of the safety and well-being of the research participant).
* No history of allergic disease i.e., a negative skin prick test(we have excluded those with allergic disease as they may have a heightened sensitivity to inhaled cough stimuli, such as the inhaled capsaicin cough challenge)
* Participants who are free from significant cardiac, gastrointestinal, hepatic, renal, haematological, neurological and psychiatric disease
* Not taking any regular medication, other than the oral contraceptive pill (we do not want any interaction with other medication that the participant may be taking i.e. we hope to measure the cough 'tussive' response in our healthy volunteers solely as a result of the effect of our compound under investigation, 2HPBCD)
* All participants must have a minimum gap of one-month from completion of a previous study, before commencement in this current study

Exclusion Criteria:

* History of respiratory disease (we have excluded those with respiratory disease so that the outcome, attenuation of the induced capsaicin cough response by intravenous 2HPBCD, is unaffected by any respiratory disease status of the participant)
* History of upper respiratory tract infection or respiratory symptoms in the preceding six weeks (as respiratory tract infections may cause cough or highly sensitize the respiratory airways to inhaled cough stimuli, such as the inhaled capsaicin cough challenge i.e. the induced cough capsaicin challenge will not be a true reflection of cough in the healthy volunteer participant)
* Evidence of a positive pregnancy test (urine beta-human chorionic gonadotrophin level) for female volunteers or female participants that are pregnant or lactating or are likely to become pregnant during the trial. Women of childbearing potential may be included in the study if, in the opinion of the investigator, they are taking adequate contraceptive precautions
* Gastrointestinal symptoms such as a recent alteration in bowel habit or new bowel symtpoms including participants with a known or suspected history of lactose intolerance (as 2HPBCD when given as an oral tablet in chronic dosing, has been shown to sometimes cause flatulence, diarrhea, soft stools and abdominal cramps)
* Participants susceptible to renal impairment from their medical history (symptoms of renal failure, medical conditions predisposing to renal impairment such as diabetes, history of recurrent urinary infection either as an adult or in childhood, history of peripheral vascular disease/stroke/coronary heart disease/hypercholestrolaemia/hyperlipidaemia), or from their medical examination (kidney size, renal bruits, peripheral upper and lower limb arterial pulses)or from their urine analysis on urine 'dipstick' (glucose, protein, blood). Any positive finding listed above will lead to exclusion of the participant from the clinical study
* Participants with an abnormal urine cytology. Any positive finding in this tests will lead to exclusion of the participant from the clinical study
* Participants who are unable to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Capsaicin Cough Challenge | 0-30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: O S Usmani, MD, PhD, Principal Investigator — Imperial College London
Locations (1):
- Asthma Lab, Royal Brompton Hospital, London, United Kingdom